CLINICAL TRIAL: NCT02355119
Title: Phase III Italian Multicenter Study Comparing the Combination of 5-fluorouracil/Folinic Acid, Oxaliplatin and Irinotecan (Folfoxiri) Versus Gemcitabine as Adjuvant Treatment for Resected Pancreatic Cancer
Brief Title: Italian Multicenter Study Comparing FOLFOXIRI Versus Gemcitabine as Adjuvant Treatment for Resected Pancreatic Cancer
Acronym: GIP-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Enrico Vasile, PI, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIP-2
Record Dates: First submitted 2015-01-20; First posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — FOLFOXIRI protocol; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine (Active Comparator): Gemcitabine 1000 mg/sqm on days 1,8,15 every 28 days
  Interventions: Drug: Gemcitabine
- FOLFOXIRI (Experimental)
  Interventions: Drug: FOLFOXIRI

INTERVENTIONS:
Drug: FOLFOXIRI — Combination of 5-Fluorouracil/Folinic Acid, Irinotecan, Oxaliplatin
  Arms: FOLFOXIRI
Drug: Gemcitabine
  Arms: Gemcitabine

SUMMARY:
Patients with resected pancreatic cancer who fulfill the selection criteria will be randomized to receive one of the two treatment arms for a period of 6 months: Gemcitabine, the standard arm, or FOLFOXIRI (the combination of 5-Fluorouracil/Folinic Acid, Oxaliplatin and Irinotecan), the experimental arm.

A total of 310 patients will be enrolled in about 50 Italian centers.

DETAILED DESCRIPTION:
Patients with resected stage I-III pancreatic cancer who fulfill the selection criteria will be randomized to receive one of the two treatment arms for a period of 6 months: Gemcitabine, the standard arm, or FOLFOXIRI (the combination of 5-Fluorouracil/Folinic Acid, Oxaliplatin and Irinotecan), the experimental arm.

A total of 310 patients will be enrolled in about 50 Italian centers. All the patients will be followed up during and after the treatment until disease progression and death or for a minimum of 60 months.

Main objective:

To show an increase in disease-free survival with an HR of 0.70 for patients enrolled into the experimental arm compared with standard arm.

Secondary objectives:

To show an increase in overall survival with an HR of 0.70 for patients enrolled into the experimental arm compared with standard arm.

To show the tolerability of the experimental treatment in this setting.

Principal inclusion criteria:

* histological diagnosis of pancreatic cancer
* surgical resection with curative intent within 10 weeks before of enrollment (stage I-III)
* absence of evidence of metastases (cM0)
* age 18-75
* ECOG performance status 0-1
* adequate bone marrow, liver and renal function
* written informed consent

Principal exclusion criteria:

* evidence of metastases
* CA19.9 higher than 2.5 x ULN (upper limit of normal range)
* precedent chemotherapy or radiotherapy
* coexisting malignancies
* relevant coexisting diseases that could contraindicate the participation to the study
* hypersensitivity/intolerance to the drugs in study
* pregnancy or breastfeeding
* neurotoxicity of grade > 1
* malabsorption syndrome

Primary end-point:

Disease-free survival, defined as the time from enrollment to the evidence of progression of disease or death.

Secondary end-points:

Overall survival, defined as the time from enrollment to the evidence of death. Toxicity, defined according to NCI-CTC

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of pancreatic cancer
* surgical resection with curative intent within 10 weeks before of enrollment (stage I-III)
* absence of evidence of metastases (cM0)
* age 18-75
* ECOG performance status 0-1
* adequate bone marrow, liver and renal function
* written informed consent

Exclusion Criteria:

* evidence of metastases
* CA19.9 higher than 2.5 x ULN (upper limit of normal range)
* precedent chemotherapy or radiotherapy
* coexisting malignancies
* relevant coexisting diseases that could contraindicate the participation to the study
* hypersensitivity/intolerance to the drugs in study
* pregnancy or breastfeeding
* neurotoxicity of grade > 1
* malabsorption syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | up to 1 year after last patient in

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 2 years after last patient in
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 28 weeks from treatment beginning

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Vasile, MD, PhD, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, PI, Italy